CLINICAL TRIAL: NCT06778590
Title: Comparison of Piezoelectric and Conventional Surgery for Germectomy of the Lower Third Molar: Assessment of Post-operative Sequelae
Brief Title: Comparison of Piezoelectric and Conventional Surgery for Germectomy of the Lower Third Molar
Acronym: Germectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amerigo Giudice (Other)
Responsible Party: Sponsor-Investigator, Amerigo Giudice, Amerigo Giudice, University Magna Graecia
Organization: University Magna Graecia (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 372/2024
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Tooth Disease; Piezoelectric Technique; Tooth Impacted; Tooth Extraction Status Nos; Tooth Avulsion; Facial Swelling; Germectomy
Keywords: third molar surgery; facial swelling; 3D facial swelling evaluation; Piezoelectric technique; tooth impacted; piezosurgery; germectomy
MeSH Terms: conditions — Tooth Diseases; Tooth, Impacted; Tooth Avulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group: Piezoelectric Surgery (Experimental): Use of piezoelectric technique in third molar germectomy procedures
  Interventions: Procedure: Piezoelectric technique in third molar germectomy
- Control group: Traditional Surgery (Active Comparator): Use of traditional technique in third molar germectomy procedures
  Interventions: Procedure: Traditional technique in third molar germectomy

INTERVENTIONS:
Procedure: Piezoelectric technique in third molar germectomy — Application of piezoelectric technique in third molar germectomy procedures
  Arms: Test group: Piezoelectric Surgery
Procedure: Traditional technique in third molar germectomy — Application of traditional technique in third molar germectomy procedures
  Arms: Control group: Traditional Surgery

SUMMARY:
The main objective of the study is to compare the effects of the piezoelectric surgery and the traditional technique on soft tissue edema in patients undergoing bilateral germectomy of mandibular third molars

DETAILED DESCRIPTION:
The main objective of the study is to compare the effects of piezoelectric surgery and the traditional technique on soft tissue edema in patients undergoing bilateral germectomy of mandibular third molars. Post-operative swelling is analyzed using a photogrammetry facial scanner (Marathon MT-4000).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 14 and 24 years, with both lower third molars in the developmental stage (with incompletely formed roots) and requiring extraction of both for prophylactic, therapeutic or strategic reasons
* Good quality of radiographic investigations (CBCT)
* Good health status

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Facial swelling qualitative analysis | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of piezosurgery in reducing facial swelling using qualitative three-dimensional analysis (measured by colorimetric variation given by the overlapping volumes)
Facial swelling quantitative analysis - volumetric differences | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of piezosurgery in reducing facial swelling using quantitative three-dimensional analysis ( volumes measured in cm3)
Facial swelling quantitative analysis - linear differences | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of piezosurgery in reducing facial swelling using quantitative three-dimensional analysis (linear differences measured in cm2)

SECONDARY OUTCOMES:
Trismus analysis | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of piezosurgery on trismus (measured in cm)
Pain analysis with Visual analogue scale (VAS) | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of piezosurgery on pain (measured by VAS-score from 0 to 10 point, with 10 as the worst outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Magna Graecia University of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No